CLINICAL TRIAL: NCT02591667
Title: Assessment of Histopathological Response to Combination Chemotherapy With Oxaliplatin, Irinotecan, Fluorouracil and Bevacizumab in Patients With Peritoneal Metastasis From Colorectal Cancer
Brief Title: Histopathological Response to FOLFOXIRI + Bevacizumab in Peritoneal Metastasis From Colorectal Cancer
Acronym: CARCINOSIS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Bachleitner-Hofmann, MD, ao.Univ.-Prof.Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-002917-30
Record Dates: First submitted 2015-10-13; First posted 2015-10-29 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Colorectal Cancer; Peritoneal Metastasis
Keywords: Colorectal cancer; Peritoneal metastasis; Neoadjuvant chemotherapy; 5-Fluorouracil; Oxaliplatin; Irinotecan; Bevacizumab; Histopathological response
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Neoadjuvant Therapy; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active treatment (Experimental): Patients will first undergo upfront staging laparoscopy with retrieval of tumor tissue for standard pathology.
  Two to 4 weeks after initial surgical exploration, patients will receive 4 cycles of FOLFOXIRI + bevacizumab, q2w. The last chemotherapy cycle will be given without bevacizumab.
  Five to 7 weeks after the last administration of bevacizumab (i.e., 3 to 5 weeks after completion of chemotherapy), patients will undergo surgery with the intent to perform complete surgical cytoreduction of all peritoneal tumor deposits. Further chemotherapy according to the currently available treatment guidelines, including intraperitoneal hyperthermic chemotherapy in patients where complete surgical cytoreduction has been achieved, will be given at the discretion of the investigator.
  Interventions: Procedure: Upfront staging laparoscopy + peritoneal biopsy; Drug: Neoadjuvant chemotherapy with FOLFOXIRI + bevacizumab; Procedure: Surgical re-exploration

INTERVENTIONS:
Procedure: Upfront staging laparoscopy + peritoneal biopsy — Upfront staging laparoscopy with biopsy of peritoneal tumor deposits, assessment of peritoneal cancer index and resectability.
Drug: Neoadjuvant chemotherapy with FOLFOXIRI + bevacizumab — Patients will receive 4 cycles of FOLFOXIRI + bevacizumab; the last cycle will be given w/o bevacizumab
  Dosage: Bevacizumab: 5 mg/kg via 30 min. IV infusion, day 1; Oxaliplatin: 85 mg/m2 via 2-hour IV infusion, day 1; Irinotecan: 165 mg/m2 via 1-hour IV infusion, day 1; Leucovorin: 200 mg/m2 via 2-hour IV infusion, day 1; 5-Fluorouracil: 3200 mg/m2 via 48-hour IV infusion, day 1;
Procedure: Surgical re-exploration — Three to 5 weeks after completion of FOLFOXIRI + bevacizumab chemotherapy, patients will undergo surgical re-exploration with the intent to perform a complete surgical cytoreduction. Further chemotherapy according to the currently available treatment guidelines, including intraperitoneal hyperthermic chemotherapy in patients where complete surgical cytoreduction has been achieved, may be given at the discretion of the investigator. Systemic chemotherapy may be started beginning 4 weeks post-surgery and after complete wound healing.

SUMMARY:
There is a paucity of data on the histopathological response of peritoneal tumor deposits from colorectal cancer to neoadjuvant chemotherapy. Particularly, no prospective assessment of chemotherapy-associated histopathological response within the peritoneum has been performed so far. Therefore, there is an urgent need to conduct a clinical trial aimed at prospectively assessing the histopathological response within the peritoneum in patients with peritoneal metastasis from colorectal cancer.

Recently, Loupakis et al. reported that the triplet regimen of 5-fluorouracil, oxaliplatin and irinotecan (FOLFOXIRI) in combination with bevacizumab significantly improved median progression-free survival in metastatic colorectal cancer patients from 9.7 to 12.1 months as compared with fluorouracil, leucovorin, and irinotecan (FOLFIRI) + bevacizumab. In view of these data, it is likely that FOLFOXIRI + bevacizumab will also lead to a significant improvement of the histopathological response within the peritoneum of patients with peritoneal metastasis from colorectal cancer (pcCRC) as compared with previous standard chemotherapy.

The investigators hypothesize that FOLFOXIRI + bevacizumab will induce a pCR or major response in peritoneal tumor deposits in >30% of patients (taking the response rate to FOLFOX- or FOLFIRI-based neoadjuvant chemotherapy from the published literature as a reference).

DETAILED DESCRIPTION:
Peritoneal carcinomatosis from colorectal cancer (pcCRC) has a dismal prognosis. In the era of 5-fluorouracil treatment and palliative surgery only, median survival ranged from 5.2 to 7.0 months. In patients with bowel obstruction due to peritoneal carcinomatosis outcome was even worse, with a median overall survival of less than 4 months and a 1-year survival rate of 17%. With the advent of modern chemotherapy regimens, survival has improved considerably. However, the presence of pcCRC is still associated with a significantly worse prognosis as compared with other manifestations of metastatic CRC (e.g. liver and/or lung metastasis). A recent retrospective analysis of 2095 patients from 2 prospective randomized trials showed that both median PFS and OS were significantly shorter for patients with pcCRC as compared with patients without pcCRC (PFS: 5.8 vs. 7.2 months, HR=1.2; 95% CI 1.1 to 1.3, p=0.001; OS: 12.7 vs. 17.6 months, HR=1.3; 95% CI 1.2 to 1.5, p<0.001).

The combination of cytoreductive surgery (CRS) with hyperthermic intraperitoneal chemotherapy (HIPEC) has led to a remarkable improvement of survival in selected patients with pcCRC as illustrated by a prospective randomized trial and several retrospective series. The concept of CRS + HIPEC has therefore recently been incorporated into national treatment guidelines and is being increasingly performed in pcCRC patients with promising long-term results. The subgroup who benefits most of this multimodal therapeutic approach are patients with limited pcCRC where a complete removal of all cancer deposits within the peritoneum can be achieved.

There is increasing evidence that the addition of neoadjuvant systemic chemotherapy to CRS + HIPEC may further improve the outcome of patients with pcCRC. Neoadjuvant chemotherapy, i.e., chemotherapy that is given upfront before CRS + HIPEC is performed, offers several possible advantages for patients: First, it can help to identify nonresponders to treatment who may be unsuitable candidates for CRS. Second, neoadjuvant chemotherapy may limit extraabdominal systemic spread of the disease. Third, upfront chemotherapy may help to reduce the extent of peritoneal metastasis, thus facilitating CRS and increasing the likelihood of a complete surgical cytoreduction.

Importantly, it has recently been shown that the efficacy of neoadjuvant chemotherapy can be easily quantified by assessing the chemotherapy-induced histopathological response within the peritoneum and that the histopathological response is an independent predictor of survival. In a retrospective analysis of 115 pcCRC patients who underwent neoadjuvant chemotherapy followed by CRS, patients were grouped into three distinct categories depending on the histopathological response to neoadjuvant chemotherapy:

1. patients with complete pathologic response (pCR; no remaining viable tumor cells in peritoneal tumor nodules),
2. patients with major response (1-49% remaining viable tumor cells) or
3. patients with minor/no response (≥50% remaining viable tumor cells).

The study was able to show that the cumulative 5-year survival rate was 75% for patients with a pCR (HR=1) as compared with 57% for patients with a major response (HR=4.91) and only 13% for patients with a minor or no response (HR=13.46) (p=0.01). Overall, approximately 30% of patients were considered to be responders to neoadjuvant chemotherapy (9.7% pCR + 20.2% major response), while about 70% of patients were considered non-responders to treatment. Treatment consisted of a FOLFOX- or FOLFIRI-based regimen in the majority of patients.

The primary objective of the study is to prospectively assess the histopathological response to neoadjuvant chemotherapy with FOLFOXIRI + bevacizumab in peritoneal tumor deposits of 30 patients with pcCRC by determining the percentage of viable tumor cells in the resected specimen after neoadjuvant chemotherapy. For patients with multiple peritoneal specimens, the median percentage of viable cells in all specimens will be used. Patients with 0-49% of viable cells will be considered as responders. The timepoint of the assessment of the primary objective will be during re-exploratory surgery/surgical cytoreduction between days 78 and 106 of the treatment phase of the study. The investigators hypothesize that there will be >30% responders after neoadjuvant chemotherapy with FOLFOXIRI + bevacizumab.

Responders will be defined as patients with pCR (0% viable tumor cells) and major response (1-49% viable tumor cells) after FOLFOXIRI + bevacizumab chemotherapy.

Non-responders will be defined as patients with minor/no response (≥50% viable tumor cells) after FOLFOXIRI + bevacizumab chemotherapy.

The following patients will also be counted as non-responders:

* Patients who do not undergo surgical re-exploration
* Patients who develop extraabdominal metastases
* Deaths before surgical re-exploration

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed carcinoma of the colon or rectum with synchronous or metachronous peritoneal metastasis.
2. Male and female patients, aged ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2.
4. Life expectancy ≥ 26 weeks.
5. Neutrophils (absolute count) ≥ 1.5 g/l.
6. Platelet count ≥ 100 g/l.
7. Hemoglobin > 9 g/dL.
8. Total bilirubin ≤ 1.8 mg/dl.
9. Aspartate aminotransferase (AST) and Alanine transaminase (ALT) ≤ 88 U/l (≤ 175 U/l if liver metastases are present).
10. Alkaline phosphatase ≤ 325 U/l (≤ 650 U/l if liver metastases are present).
11. Calculated creatinine clearance > 50 mL/min OR serum creatinine ≤ 1.5 mg/dl.
12. Proteinuria < 2+ by dipstick or urine protein <1 g by 24-hr urine collection.
13. Not pregnant or nursing.
14. Negative pregnancy test (for females of childbearing potential).
15. Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last study treatment.
16. Written informed consent.
17. General condition considered feasible for major abdominal surgery after systemic chemotherapy.
18. ≤3 liver metastases amenable to curative resection using a minor liver resection.

Exclusion Criteria:

1. Major surgical procedure or significant traumatic injury within 28 days prior to study enrolment (surgical exploration with diagnostic biopsy/sampling of peritoneal tumor deposits but without bowel resection or comparable surgical procedure is allowed).
2. History of previous cytoreductive surgery in combination with hyperthermic intraperitoneal chemotherapy.
3. Pregnancy or lactation.
4. Inability or unwillingness to comply with the protocol.
5. Evidence of current extraabdominal metastatic disease. Prior extraabdominal metastatic disease is allowed, provided that it has been curatively resected ≥6 months before study entry and that current staging shows no evidence of disease recurrence.
6. >3 liver metastases or any liver metastases not amenable to upfront curative resection using a minor liver resection.
7. Prior systemic chemotherapy completed ≤3 months before study inclusion.
8. Treatment with any other investigational agent, or participation in another clinical trial within 30 days prior to entering this study.
9. History or evidence upon physical/neurological examination of central nervous system (CNS) disease (unrelated to cancer) unless adequately treated with standard medical therapy (e.g. uncontrolled seizures).
10. Untreated brain metastases, spinal cord compression or primary brain tumors.
11. Past or current history (within the last 2 years prior to treatment start) of other malignancies except colorectal cancer (patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible).
12. Clinically significant cardiovascular disease, for example cerebrovascular accident (CVA), myocardial infarction (≤12 months before treatment start), unstable angina, New York Heart Association (NYHA) > Class II congestive heart failure (CHF), arrhythmia requiring medication, or uncontrolled hypertension.
13. Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of study enrolment.
14. Any previous venous thromboembolism > NCI Common Toxicity Criteria for Adverse Effects (CTCAE) Grade 3.
15. Prior history of hypertensive crisis or hypertensive encephalopathy.
16. Evidence of bleeding diathesis or significant coagulopathy.
17. History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or active gastrointestinal bleeding within 6 months prior to the first study treatment.
18. Known hypersensitivity to any of the study drugs.
19. Serious, non-healing wound, ulcer or bone fracture.
20. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that puts the patient at high risk for treatment-related complications.
21. Symptomatic peripheral neuropathy ≥ grade 1 according to the NCI Common Toxicity Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of viable cells within the resected peritoneal deposits after completion of neoadjuvant chemotherapy with FOLFOXIRI + bevacizumab. | at the time of surgical re-exploration (days 78 to 106)
  The percentage of viable cells within the resected specimen after completion of neoadjuvant chemotherapy will be determined. For patients with multiple peritoneal specimens, the median percentage of viable cells in all specimens will be calculated. Patients with 0-49 % of viable cells will be considered as responders.

SECONDARY OUTCOMES:
Change in the percentage of viable cells in peritoneal tumor deposits before and after completion of neoadjuvant chemotherapy. | at the time of surgical re-exploration (days 78 to 106)
  In case of multiple specimens, the change in the median percentages of viable cells in peritoneal tumor deposits between baseline and after completion of neoadjuvant chemotherapy will be compared.
Change in Peritoneal Cancer Index (PCI) between baseline and after completion of neoadjuvant chemotherapy with FOLFOXIRI + bevacizumab. | at the time of surgical re-exploration (days 78 to 106)
Change in resectability (the ability to achieve a complete surgical cytoreduction) between initial surgical exploration and surgical re-exploration after administration of combination chemotherapy with FOLFOXIRI + bevacizumab. | at the time of surgical re-exploration (days 78 to 106)
Radiologic response to combination chemotherapy with FOLFOXIRI + bevacizumab as assessed by 18F-2-fluoro-2-deoxy-D-glucose (FDG)-PET CT/MRI. | days 71 to 106
Incidence of treatment-emergent adverse events. | through study completion, an average of 12 months
Relapse-free survival (RFS) | from date of complete surgical cytoreduction until the date of first documented relapse, assessed up to 60 months
Progression-free survival (PFS) | from date of study enrolment until metastatic tumor progression or death from any cause, assessed up to 60 months
Overall survival (OS) | through study completion, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bachleitner-Hofmann, MD, Principal Investigator — Medical University of Vienna
Locations (2):
- Austria (2):
  - Medical University of Vienna, Department of Internal Medicine I, Vienna
  - Medical University of Vienna, Department of Surgery, Vienna

REFERENCES:
- [Background] Passot G, You B, Boschetti G, Fontaine J, Isaac S, Decullier E, Maurice C, Vaudoyer D, Gilly FN, Cotte E, Glehen O. Pathological response to neoadjuvant chemotherapy: a new prognosis tool for the curative management of peritoneal colorectal carcinomatosis. Ann Surg Oncol. 2014 Aug;21(8):2608-14. doi: 10.1245/s10434-014-3647-0. Epub 2014 Mar 26. PMID 24668148
- [Background] Loupakis F, Cremolini C, Masi G, Lonardi S, Zagonel V, Salvatore L, Cortesi E, Tomasello G, Ronzoni M, Spadi R, Zaniboni A, Tonini G, Buonadonna A, Amoroso D, Chiara S, Carlomagno C, Boni C, Allegrini G, Boni L, Falcone A. Initial therapy with FOLFOXIRI and bevacizumab for metastatic colorectal cancer. N Engl J Med. 2014 Oct 23;371(17):1609-18. doi: 10.1056/NEJMoa1403108. PMID 25337750
- [Background] Cremolini C, Loupakis F, Antoniotti C, Lonardi S, Masi G, Salvatore L, Cortesi E, Tomasello G, Spadi R, Zaniboni A, Tonini G, Barone C, Vitello S, Longarini R, Bonetti A, D'Amico M, Di Donato S, Granetto C, Boni L, Falcone A. Early tumor shrinkage and depth of response predict long-term outcome in metastatic colorectal cancer patients treated with first-line chemotherapy plus bevacizumab: results from phase III TRIBE trial by the Gruppo Oncologico del Nord Ovest. Ann Oncol. 2015 Jun;26(6):1188-1194. doi: 10.1093/annonc/mdv112. Epub 2015 Feb 23. PMID 25712456
- [Background] Verwaal VJ, van Ruth S, de Bree E, van Sloothen GW, van Tinteren H, Boot H, Zoetmulder FA. Randomized trial of cytoreduction and hyperthermic intraperitoneal chemotherapy versus systemic chemotherapy and palliative surgery in patients with peritoneal carcinomatosis of colorectal cancer. J Clin Oncol. 2003 Oct 15;21(20):3737-43. doi: 10.1200/JCO.2003.04.187. PMID 14551293
- [Background] Elias D, Gilly F, Boutitie F, Quenet F, Bereder JM, Mansvelt B, Lorimier G, Dube P, Glehen O. Peritoneal colorectal carcinomatosis treated with surgery and perioperative intraperitoneal chemotherapy: retrospective analysis of 523 patients from a multicentric French study. J Clin Oncol. 2010 Jan 1;28(1):63-8. doi: 10.1200/JCO.2009.23.9285. Epub 2009 Nov 16. PMID 19917863